CLINICAL TRIAL: NCT01336647
Title: An Efficacy and Safety Study of Ha44 Gel Administered Topically for the Treatment of Head Lice Infestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ha02-003
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Pediculosis
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Group A Low-Dose Ha44 Gel 0.37% w/w topically administered to head and scalp.Single application for 10 minutes.
  Interventions: Drug: Group A - Low-Dose Ha44 0.37% w/w
- Group B (Experimental): Group B High-Dose Ha44 Gel 0.74% w/w. Topically administered to hair and scalp. Single application for 10 minutes of duration.
  Interventions: Drug: Group B - High Dose Ha44 Gel 0.74% w/w
- Group C (Placebo Comparator): Group C Placebo/ vehicle Ha44 Gel. Topically administered to hair and scalp.Single application for 10 minutes of duration.
  Interventions: Drug: Group C - Placebo

INTERVENTIONS:
Drug: Group A - Low-Dose Ha44 0.37% w/w — Low Dose Ha44 Gel applied to scalp and hair for 10 minutes
  Arms: Group A
Drug: Group B - High Dose Ha44 Gel 0.74% w/w — High Dose Ha44 Gel applied to scalp and hair for 10 minutes
  Arms: Group B
Drug: Group C - Placebo — Placebo- vehicle Ha44 Gel without active ingredient applied to scalp and hair for 10 minutes
  Arms: Group C

SUMMARY:
Phase 2 study to assess the safety and effectiveness of a product to treat children and adults with head lice

ELIGIBILITY:
Inclusion Criteria:

* 2 years of age or older
* Body weight of at least 33 pounds
* Has an active head lice infestation at Day 0. An active infection is defined as at least 3 live lice for the index subject and at least 1 live louse for the other household members
* Belong to a household of no more than 6 members, except where additional household members are < 2 years of age
* Belong to a household with an eligible index subject between 2 and 12 years of age with active lice infestation
* Female subjects must be:

  * of non-childbearing potential (no history of menstrual periods, post-hysterectomy, or, post-menopausal for at least 2 years) OR,
  * if of childbearing potential, must have a negative urine pregnancy test prior to treatment and agree to use a highly effective method of contraception from Day 0 through the Day 14 visit.

Exclusion Criteria:

* Had treatment for head lice within 14 days prior to Day 0
* Has a household member(s) who is infested with lice but is not willing or not eligible for enrollment
* Has a condition or illness that, in the opinion of the Investigator, may interfere with the study results
* Has an electrocardiographic abnormality, renal disease or impaired renal function, dermatological disease on the face, scalp, ears or neck, or active ophthalmological disease, moderate or severe scleral injection with conjunctival erythema or purulent discharge or allergic or perennial rhinitis requiring chronic treatment
* Has been using hormonal contraception for less than 3 months or is pregnant or lactating
* Has received systemic corticosteroids within 7 days prior to Day 0 or planned while on study
* Receiving systemic or topical medication, which in the opinion of the Investigator, may interfere with the study results
* Has received an investigational agent within 30 days prior to Day 0

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Restrepo, Principal Investigator — Universal Biopharma Reserach Inc.; Lydie Hazan, Principal Investigator — Axis Clinical Trials
Locations (2):
- United States (2):
  - Universal BioPharma Research Institute, Inc., Dinuba, California
  - Axis Clinical Trials, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Ha 44 Gel: Low-Dose Ha44 Gel 0.37%, it was administered topically for 10 minutes as a single dose.
- High-Dose Ha44: High-Dose Ha44 Gel 0.74% it was administered topically for 10 minutes as a single dose
- Vehicle: Vehicle Ha44 Gel with no active incident it was administered topically for 10 minutes as a single dose.
Period: Overall Study
Arm/Group | Low Dose Ha 44 Gel | High-Dose Ha44 | Vehicle
Started | 46 | 49 | 47
Completed | 42 | 48 | 44
Not Completed | 4 | 1 | 3
Not completed — Lost to Follow-up | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Ha44 Gel: Low-Dose Ha44 0.37% Gel, topically administered to hair and scalp for 10 minutes
- High-Dose Ha44: High-Dose Ha44 0.74% Gel, topically administered to hair and scalp for 10 minutes
- Vehicle: Vehicle Gel without active ingredient of Ha44.
- Total: Total of all reporting groups
Arm/Group | Low Dose Ha44 Gel | High-Dose Ha44 | Vehicle | Total
Number analyzed (Participants) | 46 | 49 | 47 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38 | 35 | 30 | 103
  Between 18 and 65 years | 8 | 14 | 17 | 39
  >=65 years | 0 | 0 | 0 | 0
Age, Customized [Mean (Standard Deviation); unit: years] | 13.7 (10.5) | 15.3 (11.3) | 17.3 (13.3) | 15.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 44 | 128
  Male | 4 | 7 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Lice Free at All Follow-up Visits (Day 1, 7 and 14) Through the Day 14 Visit
Time Frame: Follow up visit at days 1, 7 and 14 days
Population: Intent to Treat
Measure: Number; unit: participants
Groups:
- Low Dose Ha44: Ha44 0.37% Gel administered topically to hair and scalp for 10 minutes.
- Hig Dose Ha44: Ha44 0.74% Gel administered topically to hair and scalp for 10 minutes.
- Vehicle: Vehicle Gel without active ingredient administered topically to hair and scalp for 10 minutes.
Arm/Group | Low Dose Ha44 | Hig Dose Ha44 | Vehicle
Number analyzed (Participants) | 46 | 49 | 47
participants | 31 | 42 | 11
Statistical Analysis 1: Comparison: Low Dose Ha44 vs Hig Dose Ha44 vs Vehicle; Null hypothesis; 80% power and 0.025 two-sided level of significance for each pairwise active vs. vehicle comparison; Test type: Non-Inferiority or Equivalence — The primary efficacy endpoint was responder rate calculated based on the percentage of subjects who were lice free at all follow-up visits (Days 1, 7 and 14). Because the number of responders and non-responders in the family size>= 5 household members was less than five in at least one of the treatment arms, (Table 14.2.1.5), Fisher's Exact test was used to compare treatment arms, instead of the CMH test; p < 0.001, Fisher Exact; The assessment of statistical significance will be done using Hochberg's modified Bonferroni test

2. Secondary Outcome: Safety and Tolerability of Ha44 Gel
Description: The number of subjects with Treatment emergent AEs (TEAEs) related to the study medication will be reported by treatment group.
Time Frame: From treatment to last visit of the study at 14 days
Population: All subjects who participated
Measure: Number; unit: participants with treatment related AEs
Groups:
- Low Dose Ha44: Low-Dose Ha44 0.37% Gel, administered topically to hair and scalp for 10 minutes.
- High Dose Ha44: High-Dose Ha44 0.74% Gel administered topically to hair and scalp for 10 minutes.
Arm/Group | Low Dose Ha44 | High Dose Ha44 | Vehicle
Number analyzed (Participants) | 46 | 49 | 47
participants with treatment related AEs | 5 | 8 | 13

ADVERSE EVENTS:
Time Frame: 14 days
Groups:
- Low Dose Ha44 Gel: Low-Dose Ha44 0.37% Gel, administered topically to hair and scalp for 10 minutes.
- High Dose Ha44 Gel: High-Dose Ha44 0.74% Gel, administered topically to hair and scalp for 10 minutes.
Arm/Group | Low Dose Ha44 Gel | High Dose Ha44 Gel | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/49 | 0/47
Other Adverse Events (participants affected / at risk) | 11/46 | 2/49 | 20/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Ha44 Gel (N=46) | High Dose Ha44 Gel (N=49) | Vehicle (N=47)
pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2) | 18 (18)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less